CLINICAL TRIAL: NCT01345721
Title: A Phase IIIb, Open-Label, Controlled, Multi-Center Study to Evaluate the Persistence Of Antibody Responses Among Children Who Previously Received Novartis MenACWY Conjugate Vaccine or Meningococcal C Conjugate Vaccine
Brief Title: Persistence Of Antibody Responses Among Children Who Previously Received Novartis MenACWY Conjugate Vaccine or Meningococcal C Conjugate Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V59P22E1
Record Dates: First submitted 2011-04-29; First posted 2011-05-02 (Estimated); Results first posted 2013-10-18 (Estimated); Last update posted 2018-06-18 (Actual); Status verified 2018-05

CONDITIONS: Meningococcal Disease
Keywords: Meningococcal; ACWY; Conjugate Vaccine; Meningitis; Toddlers; Children; Persistence; Boost
MeSH Terms: conditions — Meningococcal Infections; Meningitis | interventions — MenACWY-CRM vaccine

ARMS (3):
- MenACWY (2 primary + 1 booster dose) (Experimental): Subjects who had previously received two primary doses of MenACWY-CRM vaccine (at 6-8 months and 12 months of age) in parent study, were administered one booster dose of the same vaccine in this extension study.
  Interventions: Biological: MenACWY-CRM
- MenACWY (1 primary + 1 booster dose) (Experimental): Subjects who had previously received one primary dose of MenACWY-CRM vaccine (at 12 months of age) in parent study, were administered one booster dose of the same vaccine in this extension study.
  Interventions: Biological: MenACWY-CRM
- MenC (1 primary dose)+MenACWY (1 booster dose) (Experimental): Subjects who had previously received one primary dose of the comparator MenC vaccine (at 12 months of age) in parent study, were administered one booster dose MenACWY-CRM vaccine in this extension study.
  Interventions: Biological: MenACWY-CRM

INTERVENTIONS:
Biological: MenACWY-CRM

SUMMARY:
The primary purpose of this study is to evaluate the persistence of bactericidal antibodies in children of approximately 22 to 45 months of age previously enrolled in the V59P22 study (NCT00667602) who received Novartis MenACWY Conjugate Vaccine or Meningococcal C Conjugate Vaccine. This is measured by percentage of subjects with human Serum Bactericidal Assay (hSBA) titers ≥ 1:8 directed against Neisseria meningitidis serogroups A, C, W-135, and Y. In addition the response one month post an additional dose of Novartis MenACWY will be measured by percentage of subjects with hSBA titers ≥ 1:8 and GMTs.

ELIGIBILITY:
Inclusion Criteria:

Children eligible to be enrolled in the study were those

* whose parents provide written informed consent;
* were in generally good health based on the clinical judgment of the investigators;
* subjects were 22-45 months of age at the time of enrollment into V59P22E1;
* subject who had participated in the parent V59P22 study.

Exclusion Criteria:

Main exclusion criteria:

* Subjects with serious, acute, or chronic illnesses
* Subjects who had received any other licensed vaccines within 28 days (Exception: Influenza vaccine was allowed up to 14 days prior to and no less than 14 days after the study immunization) prior to enrolment and any study visit
* Subjects who had received any Meningococcal vaccine since the study dose of MenACWY or Men C at 12 months of age in V59P22 trial.

Ages: 22 Months to 45 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 205 (Actual)
Dates: Start 2011-05; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (11):
- Germany (11):
  - Dr. Johannes Kandzora and Dr. Kathrin Kandzora, Am Teich 11, Neumuenster
  - Bogda-Maria Kniese,, Boyneburgstr 7, Eschwege
  - Dr Goertz Martin Kimmig, GroBbottwarer Str 47, Oberstenfeld
  - Dr med Walter Otto, Heinrichstrasse 16 A, Fulda
  - Dr med Kerstin Pscherer, Hellersdorfer Str 237, Berlin
  - Dr Renate Mangelsdorf-Taxis, Kirchstrasse 2, Bonnigheim
  - Dr. Christoph Wittermann, Murnauer Str 3, Weilheim
  - Ute Jessat, Rathausstr 6, Gluecksburg
  - Dr med Luise Schroeter, Schoenwalder Str 28, Berlin
  - Dr med Ulrich Pfletschinger, Stuttgarter Strasse 74, Stuttgart Feuerbach
  - Dr Lothar Maurer, Welschgasse 39, Frankenthal

REFERENCES:
- [Derived] Giuliani MM, Biolchi A, Keshavan P, Moriondo M, Tomei S, Santini L, Mori E, Brozzi A, Bodini M, Nieddu F, Ricci S, Mzolo T, Costantini M, Azzari C, Pellegrini M. Bactericidal antibodies against hypervirulent Neisseria meningitidis C field strains following MenC-CRM or MenACWY-CRM priming and MenACWY-CRM booster in children. Hum Vaccin Immunother. 2021 May 4;17(5):1442-1449. doi: 10.1080/21645515.2020.1833578. Epub 2020 Dec 16. PMID 33325757

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects for this extension study were enrolled from only sites in Germany that participated in the parent study.
Pre-assignment Details: All enrolled subjects were included in the trial.
Groups:
- MenACWY (2 Primary + 1 Booster Dose): Subjects, who had previously received two primary doses of MenACWY-CRM vaccine (at 6-8 months and 12 months of age) in parent study, were administered one booster dose of the same vaccine in this extension study.
- MenACWY (1 Primary + 1 Booster Dose): Subjects, who had previously received one primary dose of MenACWY-CRM vaccine (at 12 months of age) in parent study, were administered one booster dose of the same vaccine in this extension study.
- MenC (1 Primary Dose) + MenACWY (1 Booster Dose): Subjects, who had previously received one primary dose of the comparator MenC vaccine (at 12 months of age) in parent study, were administered one booster dose MenACWY-CRM vaccine in this extension study.
Period: Overall Study
Arm/Group | MenACWY (2 Primary + 1 Booster Dose) | MenACWY (1 Primary + 1 Booster Dose) | MenC (1 Primary Dose) + MenACWY (1 Booster Dose)
Started | 74 | 66 | 65
Completed | 74 | 66 | 65
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- MenACWY (2 Primary +1 Booster Dose): Subjects, who had previously received two primary doses of MenACWY-CRM vaccine (at 6-8 months and 12 months of age) in parent study, were administered one booster dose of the same vaccine in this extension study.
- MenC (1 Primary Dose) +MenACWY (1 Booster Dose): Subjects, who had previously received one primary dose of the comparator MenC vaccine (at 12 months of age) in parent study, were administered one booster dose MenACWY-CRM vaccine in this extension study.
- Total: Total of all reporting groups
Arm/Group | MenACWY (2 Primary +1 Booster Dose) | MenACWY (1 Primary + 1 Booster Dose) | MenC (1 Primary Dose) +MenACWY (1 Booster Dose) | Total
Number analyzed (Participants) | 74 | 66 | 65 | 205
Age, Continuous [Mean (Standard Deviation); unit: months] | 36.7 (5.3) | 37.4 (5.6) | 37.9 (5.3) | 37.3 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 30 | 37 | 101
  Male | 40 | 36 | 28 | 104

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Persisting Serum Bactericidal Antibody Titers ≥1:8, Upto 13-33 Months After Primary Vaccination With Either MenACWY-CRM or MenC Vaccine
Description: The percentage of subjects with persisting serum bactericidal antibody (hSBA)titers ≥1:8 against Neisseria meningitidis serogroups A,C,W,Y, 13-33 months after receiving either one or two doses of MenACWY-CRM conjugate vaccine or one dose of MenC vaccine in parent study, is reported.
  The functional bactericidal antibodies response against N. meningitidis serogroups was measured with the serum bactericidal assay using human complement (hSBA)
Time Frame: From 13-33 months post last vaccination in parent study (V59P22)
Population: The analysis was done on the per-protocol persistence dataset i.e all enrolled subjects who provided evaluable serum samples at day 1 of the study and had no major protocol violation as defined prior to the end of the study.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | MenACWY (2 Primary + 1 Booster Dose) | MenACWY (1 Primary + 1 Booster Dose) | MenC (1 Primary Dose) +MenACWY (1 Booster Dose)
Number analyzed (Participants) | 52 | 41 | 43
Percentages of subjects
  13-33 months persistence (Serogroup A) | 13 [6 to 26] | 7 [2 to 20] | 0 [0 to 8]
  13-33 months persistence (Serogroup C)(N=52,40,42) | 27 [16 to 41] | 25 [13 to 41] | 36 [22 to 52]
  13-33 months persistence (Serogroup W-135) | 50 [36 to 64] | 63 [47 to 78] | 12 [4 to 25]
  13-33 months persistence (Serogroup Y) | 40 [27 to 55] | 39 [24 to 55] | 19 [8 to 33]

2. Secondary Outcome: Persisting Geometric Mean Titers in Children, 13-33 Months After Primary Vaccination With Either MenACWY-CRM or MenC Vaccine
Description: The persisting serum bactericidal antibody titers in children, 13-33 months after receiving either one or two doses of MenACWY-CRM vaccine or one dose of Men C vaccine in the parent study, are reported as GMTs against N. meningitidis serogroups A,C, W,Y
Time Frame: From 13-33 months post last vaccination in parent study (V59P22)
Population: The analysis was done on the per-protocol persistence dataset.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | MenACWY (2 Primary + 1 Booster Dose) | MenACWY (1 Primary + 1 Booster Dose) | MenC (1 Primary Dose) + MenACWY (1 Booster Dose)
Number analyzed (Participants) | 52 | 41 | 43
Titers
  13-33 months persistence (Serogroup A) | 2.82 [2.36 to 3.37] | 2.52 [2.05 to 3.08] | 2 [1.64 to 2.43]
  13-33 months persistence (Serogroup C) N=52,40 | 3.94 [2.92 to 5.3] | 3.93 [2.79 to 5.53] | 4.94 [3.55 to 6.86]
  13-33 months persistence (Serogroup W-135) | 9.36 [6.31 to 14] | 12 [7.53 to 18] | 2.81 [1.82 to 4.32]
  13-33 months persistence (Serogroup Y) | 6.79 [4.87 to 9.47] | 6.03 [4.14 to 8.78] | 2.99 [2.08 to 4.3]

3. Primary Outcome: Percentage of Subjects With Serum Bactericidal Antibody Titers ≥1:8, One Month After MenACWY-CRM Booster Vaccination
Description: The serum antibody response following a booster dose of MenACWY-CRM conjugate vaccine in children, who had previously received either one or two doses of the same vaccine in the parent study, is reported as percentage of subjects with hSBA titers ≥1:8 against N. meningitidis serogroups A,C,W,Y.
Time Frame: 1 month post booster
Population: The analysis was done on the per-protocol dataset i.e All enrolled subjects who correctly received the vaccine, provided evaluable serum samples at the relevant time points (Day 28),and had no major protocol violation as defined prior to the end of the study.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | MenACWY (2 Primary + 1 Booster Dose) | MenACWY (1 Primary + 1 Booster Dose)
Number analyzed (Participants) | 52 | 41
Percentages of subjects
  Pre-booster (Serogroup A) | 13 [6 to 26] | 7 [2 to 20]
  1 month post booster (Serogroup A) | 96 [87 to 100] | 98 [87 to 100]
  Pre-booster (Serogroup C) N=52,40 | 27 [16 to 41] | 25 [13 to 41]
  1 month post booster (Serogroup C) N=52,40 | 100 [93 to 100] | 100 [91 to 100]
  Pre-booster (Serogroup W-135) | 50 [36 to 64] | 63 [47 to 78]
  1 month post booster (Serogroup W-135) | 100 [93 to 100] | 100 [91 to 100]
  Pre-booster (Serogroup Y) | 40 [27 to 55] | 39 [24 to 55]
  1 month post booster (Serogroup Y) | 100 [93 to 100] | 100 [91 to 100]

4. Primary Outcome: Geometric Mean Titers in Children,One Month After MenACWY-CRM Booster Vaccination
Description: The serum antibody titers following a booster dose of MenACWY-CRM conjugate vaccine in children, who had previously received either one or two doses of the same vaccine in the parent study, are reported as geometric mean titers (GMTs) against N. meningitidis serogroups A,C, W,Y.
Time Frame: 1 month post booster vaccination
Population: The analysis was done on the per-protocol dataset.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | MenACWY (2 Primary + 1 Booster Dose) | MenACWY (1 Primary + 1 Booster Dose)
Number analyzed (Participants) | 52 | 41
Titers
  Pre-booster (Serogroup A) | 2.82 [2.35 to 3.38] | 2.52 [2.05 to 3.09]
  1 month post booster (Serogroup A) | 182 [118 to 281] | 214 [131 to 350]
  Pre-booster (Serogroup C) N=52,40 | 3.92 [2.92 to 5.26] | 3.91 [2.79 to 5.48]
  1 month post booster (Serogroup C) N=52,40 | 541 [399 to 733] | 968 [682 to 1372]
  Pre-booster (Serogroup W-135) | 9.37 [6.3 to 14] | 12 [7.51 to 18]
  1 month post booster (Serogroup W-135) | 799 [564 to 1133] | 1267 [854 to 1879]
  Pre-booster (Serogroup Y) | 6.79 [4.86 to 9.5] | 6.04 [4.13 to 8.82]
  1 month post booster (Serogroup Y) | 650 [448 to 941] | 676 [444 to 1027]

5. Primary Outcome: Percentage of Subjects (Who Had Previously Received MenC Vaccine) With Serum Bactericidal Antibody Titers ≥ 1:8, After One Dose of MenACWY-CRM Vaccination
Description: The serum antibody response following a dose of MenACWY-CRM conjugate vaccine in children, who had previously received one dose of MenC vaccine in the parent study, is reported as percentage of subjects with hSBA titers ≥1:8 against N. meningitidis serogroups A,C, W,Y
Time Frame: 1 month after vaccination
Population: The analysis was done on the per-protocol dataset.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | MenC (1 Primary Dose) +MenACWY (1 Booster Dose)
Number analyzed (Participants) | 41
Percentages of subjects
  Pre-vaccination (Serogroup A) | 0 [0 to 9]
  1 month post vaccination (Serogroup A) | 61 [45 to 76]
  Pre-vaccination (Serogroup C) N=39 | 36 [21 to 53]
  1 month post vaccination (Serogroup C) N=39 | 100 [91 to 100]
  Pre-vaccination (Serogroup W-135) | 12 [4 to 26]
  1 month post vaccination (Serogroup W-135) | 95 [83 to 99]
  Pre-vaccination (Serogroup Y) | 20 [9 to 35]
  1 month post vaccination (Serogroup Y) | 95 [83 to 99]

6. Primary Outcome: Geometric Mean Titers in Children (Who Previously Received MenC Vaccine) One Month After One Dose of MenACWY-CRM Vaccine
Description: The serum antibody titers following one dose of MenACWY-CRM conjugate vaccine in children, who had previously received one dose of MenC vaccine in the parent study, are reported as GMTs against N. meningitidis serogroups A,C,W,Y
Time Frame: 1 month post vaccination
Population: The analysis was done on the per-protocol dataset.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | MenC (1 Primary Dose) +MenACWY (1 Booster Dose)
Number analyzed (Participants) | 41
Titers
  Pre-vaccination (Serogroup A) | 2 [1.63 to 2.45]
  1 month post vaccination (Serogroup A) | 20 [12 to 32]
  Pre-vaccination (Serogroup C) N=39 | 4.83 [3.44 to 6.77]
  1 month post vaccination (Serogroup C) N=39 | 1530 [1077 to 2173]
  Pre-vaccination (Serogroup W-135) | 2.82 [1.81 to 4.39]
  1 month post vaccination (Serogroup W-135) | 54 [37 to 80]
  Pre-vaccination (Serogroup Y) | 3.05 [2.09 to 4.44]
  1 month post vaccination (Serogroup Y) | 54 [35 to 81]

7. Secondary Outcome: Percentage of Subjects With Serum Bactericidal Titers ≥1:8, Who Previously Received 1 Primary Dose of Either MenACWY-CRM or Men C Vaccine
Description: Comparison of serum antibody responses following one dose of MenACWY-CRM conjugate vaccine in children, who had previously received either one dose of the same vaccine or one dose of Men C vaccine in the parent study, is reported as percentage of subjects with hSBA titers ≥1:8 against N. meningitidis serogroups A,C,W,Y
Time Frame: 1 month post vaccination
Population: The analysis was done on the per-protocol dataset
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | MenACWY (1 Primary + 1 Booster Dose) | MenC (1 Primary Dose) +MenACWY (1 Booster Dose)
Number analyzed (Participants) | 41 | 41
Percentages of subjects
  hSBA ≥1:8(Serogroup A) | 98 [87 to 100] | 61 [45 to 76]
  hSBA ≥1:8 (Serogroup C) N=40,39 | 100 [91 to 100] | 100 [91 to 100]
  hSBA ≥1:8(Serogroup W-135) | 100 [91 to 100] | 95 [83 to 99]
  hSBA ≥1:8 (Serogroup Y) | 100 [91 to 100] | 95 [83 to 99]

8. Secondary Outcome: Geometric Mean Titers Following One Dose of MenACWY-CRM Vaccine in Children Who Previously Received 1 Primary Dose of Either MenACWY-CRM or Men C Vaccine
Description: Comparison of serum antibody titers following a one dose of MenACWY-CRM conjugate vaccine in children, who had previously received either one dose of the same vaccine or one dose of MenC vaccine in the parent study, are reported as GMTs against N. meningitidis serogroups A,C, W,Y
Time Frame: 1 month post vaccination
Population: The analysis was done on the per-protocol dataset
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | MenACWY (1 Primary + 1 Booster Dose) | MenC (1 Primary Dose) +MenACWY (1 Booster Dose)
Number analyzed (Participants) | 41 | 41
Titers
  1 month post vaccination (Serogroup A) | 214 [131 to 350] | 20 [12 to 32]
  1 month post vaccination (Serogroup C) N=40,39 | 968 [682 to 1372] | 1530 [1077 to 2173]
  1 month post vaccination (Serogroup W-135) | 1267 [854 to 1879] | 54 [37 to 80]
  1 month post vaccination (Serogroup Y) | 676 [444 to 1027] | 54 [35 to 81]

9. Secondary Outcome: Number of Children Reporting Solicited Local and Systemic Adverse Events (AEs) After MenACWY-CRM Vaccination
Description: The safety and tolerability of MenACWY-CRM vaccine in children (who had previously received either one or two doses of MenACWY-CRM vaccine or one dose of MenC vaccine in the parent study) is assessed in terms of number of subjects reporting solicited local and systemic AEs after MenACWY-CRM vaccine.
Time Frame: Day 1-7 after vaccination
Population: The analysis was done on the safety dataset i.e all subjects who received the study vaccine and provided some post-vaccination safety data
Measure: Number; unit: Participants
Arm/Group | MenACWY (2 Primary + 1 Booster Dose) | MenACWY (1 Primary + 1 Booster Dose) | MenC (1 Primary Dose) + MenACWY (1 Booster Dose)
Number analyzed (Participants) | 53 | 44 | 43
Participants
  Any Solicited Local | 33 | 30 | 30
  Injection site pain | 10 | 15 | 13
  Injection site erythema | 14 | 17 | 15
  Injection site induration | 6 | 8 | 7
  Any Solicited Systemic | 28 | 18 | 25
  Arthralgia | 1 | 5 | 4
  Headache | 5 | 6 | 1
  Vomiting | 0 | 2 | 1
  Change in eating habits | 6 | 8 | 6
  Rash | 0 | 2 | 1
  Sleepiness | 10 | 13 | 10
  Fever (≥38°C) | 8 | 7 | 7
  Any other | 5 | 7 | 5
  Stayed at home | 4 | 5 | 2
  Analgesic Antipyretic Medication Used | 4 | 6 | 5
  Temperature (≥40°C) (N= 52,41,41) | 0 | 0 | 2

10. Secondary Outcome: Number of Children Reporting Unsolicited Adverse Events After MenACWY-CRM Vaccination
Description: The safety of MenACWY-CRM vaccine in children (who had previously received either one or two doses of MenACWY-CRM vaccine or one dose of MenC vaccine in the parent study) is assessed in terms of number of subjects reporting any unsolicited AEs (day 1 to day 7); serious AEs and AEs necessitating medical attention/or premature withdrawal (day 1 to day 28) after MenACWY-CRM vaccine.
Time Frame: Day 1-28 after vaccination
Population: The analysis was done on the safety dataset.
Measure: Number; unit: Participants
Arm/Group | MenACWY (2 Primary + 1 Booster Dose) | MenACWY (1 Primary + 1 Booster Dose) | MenC (1 Primary Dose) + MenACWY (1 Booster Dose)
Number analyzed (Participants) | 53 | 44 | 43
Participants
  Any AE | 11 | 10 | 9
  At least possibly related AEs | 0 | 2 | 1
  Serious AE | 0 | 0 | 0
  AEs leading to premature withdrawal | 0 | 0 | 0
  Deaths | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Solicited and unsolicited AEs were collected from Day 1-7 after vaccination. SAEs and AEs necessitating medical attention/premature withdrawal were collected from Day 1-28.
Description: Due to non-compliance with protocol, data from one site was excluded in the parent study and subsequently from this extension study.Thus the number of subjects analyzed for safety differ from enrolled population.
Arm/Group | MenACWY (2 Primary + 1 Booster Dose) | MenACWY (1 Primary + 1 Booster Dose) | MenC (1 Primary Dose) + MenACWY (1 Booster Dose)
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/44 | 0/43
Other Adverse Events (participants affected / at risk) | 33/53 | 31/44 | 30/43
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MenACWY (2 Primary + 1 Booster Dose) (N=53) | MenACWY (1 Primary + 1 Booster Dose) (N=44) | MenC (1 Primary Dose) + MenACWY (1 Booster Dose) (N=43)
Diarrhoea (Gastrointestinal disorders) | 4 | 2 | 8
Injection site erythema (General disorders) | 14 | 17 | 15
Injection site induration (General disorders) | 6 | 8 | 7
Injection site pain (General disorders) | 10 | 15 | 13
Irritability (General disorders) | 12 | 8 | 14
Pyrexia (General disorders) | 8 | 8 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 5 | 4
Headache (Nervous system disorders) | 5 | 6 | 1
Somnolence (Nervous system disorders) | 10 | 13 | 10
Eating disorder (Psychiatric disorders) | 6 | 8 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days